CLINICAL TRIAL: NCT04451200
Title: Sequential and Personalized Pharmacokinetic-guided Busulfan Administration in the Frame of the Conditiong Regimen for Allogeneic Haematopoietic Stem Cell Transplantation in Patients With Malignant Hemopathies Ineligible for the Standard Myeloablative Conditioning
Brief Title: Sequential and Personalized PK-guided Busulfan Administration in the Frame of the Conditiong Regimen for Allo-HSCT in Patients With Malignant Hemopathies Ineligible for the Standard Myeloablative Conditioning
Acronym: BUSEQ
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUSEQ-IPC 2020-006
Record Dates: First submitted 2020-06-03; First posted 2020-06-30 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Acute Leukemia; Mielodysplasic Syndrome; Myeloproliferative Neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- busulfan treatment (Experimental): Personalized BU administration
  Interventions: Drug: Busulfan Injection

INTERVENTIONS:
Drug: Busulfan Injection — injections doses will be personalized by PK at days -7 and -4

SUMMARY:
Because the anti-leukemic activity of busulfan, this dug is largely used in graft conditioning but in elderly and/or cormobid patienth an excess of toxicity is observed. This study focus on the possibility of significanty reducing this toxicity by customizing the doses of busulfan to individual PK parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient up to 65 years old
* Acute leukemia, myelodysplastic syndrome or myeloproliferative neoplasia eligible for an allogeneic transplant
* Chemosensitive disease, in complete or partial or stable remission
* Allograft from an identical HLA related donor, Haplo-identical or unrelated (HLA compatibility from 8/10 to 10/10 according to HLA-A, -B, -C, -DR, -DQ allelics)
* Signed consent to participate

  -. Affiliation to a social security regimen or beneficiary of this regimen
* Patient not eligible for standard myeloablative conditioning due to age> = 45 years and / or the presence of an HCT-CI comorbidity score> = 3

Exclusion Criteria:

* Pregnant woman, without effective contraception or breastfeeding
* Person in emergency situation, patient deprived of liberty or placed under the authority of a tutor,
* Impossibility of undergoing medical follow-up of the trial for geographic, social or psychological reasons
* Contraindications to performing an allogeneic transplant
* Previous allograft
* Placental blood allograft

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
non-relapse mortality evaluation | 100 days post graft
  non-relapse mortality evaluation

SECONDARY OUTCOMES:
incidence of grade 3 or 4 toxicities | 1 month
  To evaluate toxicities linked to sequential bususlfan administration
graft taking after sequential busulfan conditioning | day 30 and day 100 post graft
  incidence of hematological reconstituation
incidence of transfusion needs for red blood cells | day 30 post graft
  number of transfusions after graft
incidence of transfusion needs for red blood cells | day 60 post graft
  number of transfusions after graft
incidence in graft taking after sequential busulfan conditioning | day 100 post graft
  Lymphocyte chimerism
anti-tumoral efficacy of sequential busulfan conditioning: incidence of acute GVH | 1 year
  incidence of acute GVH
anti-tumoral efficacy of sequential busulfan conditioning: incidence of acute GVH | 5 years
  incidence of acute GVH
the anti-tumoral efficacy of sequential busulfan conditioning: incidence of chronic GVH | 1 and 5 years
  incidence of chronic GVH
the anti-tumoral efficacy of sequential busulfan conditioning: incidence of chronic GVH | 1 year
  incidence of chronic GVH
anti-tumoral efficacy of sequential busulfan conditioning: progression-free survival | 5 years
  progression-free survival
anti-tumoral efficacy of sequential busulfan conditioning: progression-free survival | 1 year
  overall survival
anti-tumoral efficacy of sequential busulfan conditioning: progression-free survival | 5 years
  overall survival
anti-tumoral efficacy of sequential busulfan conditioning: Incidence of relapse | 1 year
  Incidence of relapse
Differences between the theoretical target AUC and the measured a posteriori | 1 month
  To study the pharmacokinetics of the sequential administration of busulfan

IPD SHARING:
Plan to Share IPD: No